CLINICAL TRIAL: NCT06403813
Title: Testing the Effectiveness of a Digital Adolescent Behavioral Health Screening, Literacy, and Low-Intensity Intervention for Common Adolescent Mental Health Problems in Kenya
Brief Title: Adolescent Digital Mental Health-Kenya Effectiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-01092; 5R21MH124149 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Mental Disorder in Adolescence
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The Kenyan study site personnel who carry out Time 2 family data collection will be masked to intervention conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Sham Comparator): Participating schools will be randomly assigned to one of the 4 study arms. Neither the parent or adolescents in the control schools will receive the intervention. Families from the control schools will be given the option to use any other version of Toolkit after completion of the Time 2 post-intervention data collection.
  Interventions: Other: Control Tooklit
- mSELY-A intervention (Experimental): Participating schools will be randomly assigned to one of the 4 study arms. Only the adolescents from the mSELY-A-alone schools will receive the mSELY-A intervention. Families from these mSELY-A-alone schools will be given the option to use any other version of Toolkit after completion of the Time 2 post-intervention data collection.
  Interventions: Behavioral: mHealth Toolkit for Screening & Empowering Lives of Youth (mSELY-A) for Adolescents
- mSELY-P intervention (Experimental): Participating schools will be randomly assigned to one of the 4 study arms. Only the parents from the mSELY-P-alone schools will receive the mSELY-P intervention. Families from these mSELY-P-alone schools will be given the option to use any other version of Toolkit after completion of the Time 2 post-intervention data collection.
  Interventions: Behavioral: mHealth Toolkit for Screening & Empowering Lives of Youth (mSELY-P) for Parents
- mSELY-A and mSELY-P intervention (Experimental): Participating schools will be randomly assigned to one of the 4 study arms. Both parent and adolescent participants from the mSELY-A+P intervention schools will receive the mSELY-A and mSELY-P intervention.
  Interventions: Behavioral: mHealth Toolkit for Screening & Empowering Lives of Youth (mSELY-A) for Adolescents; Behavioral: mHealth Toolkit for Screening & Empowering Lives of Youth (mSELY-P) for Parents

INTERVENTIONS:
Behavioral: mHealth Toolkit for Screening & Empowering Lives of Youth (mSELY-A) for Adolescents — mSELY is a preventive intervention tool to be used by adolescents and/or their parents as a self-help support modality. The mSELY-A is designed for adolescents to self-evaluate and manage psychological wellbeing/mental health needs, as well as to gain resources and access and connect with adolescent peers.The mSELY integrates 4 key mental health service functions: i) screening for common mental health problems (anxiety, depression, conduct problems) in adolescents and social-cognitive-behavioral-environmental risks in multiple domains; ii) a strength and weakness profile for adolescents' behaviors (to promote self-awareness); iii) tailored mental health literacy and promotion strategies, and iv) tailored referral resources (ii to iv are to be generated from the i screening results).
  Arms: mSELY-A and mSELY-P intervention; mSELY-A intervention
Behavioral: mHealth Toolkit for Screening & Empowering Lives of Youth (mSELY-P) for Parents — mSELY is a preventive intervention tool to be used by adolescents and/or their parents as a self-help support modality. The mSELY-P is designed for parents to self-evaluate their adolescent's development and mental health, gain awareness about their adolescent's mental health status, and learn strategies and resources to support adolescents' mental health. The mSELY integrates 4 key mental health service functions: i) screening for common mental health problems (anxiety, depression, conduct problems) in adolescents and social-cognitive-behavioral-environmental risks in multiple domains; ii) a strength and weakness profile for adolescents' behaviors (to promote self-awareness); iii) tailored mental health literacy and promotion strategies, and iv) tailored referral resources (ii to iv are to be generated from the i screening results).
  Arms: mSELY-A and mSELY-P intervention; mSELY-P intervention
Other: Control Tooklit — The toolkit will have the same screening questions, with information, but without any decision support functions.
  Arms: Control

SUMMARY:
This study seeks to respond to the growing burden of adolescent mental health disorders and urgent preventive service needs in Kenya by studying the effectiveness of a digital health intervention- mobile health (mHealth) Toolkit for Screening & Empowering Lives of Youth (mSELY)-that has demonstrated feasibility from our prior pilot study. The investigators will build on this work and examine two versions of mSELY. The mSELY-A is designed for adolescents to self-evaluate and manage psychological wellbeing/mental health needs, as well as to gain resources and access and connect with adolescent peers. The mSELY-P is designed for parents to self-evaluate their adolescent's development and mental health, gain awareness about their adolescent's mental health status, and learn strategies and resources to support adolescents' mental health. Both versions provide screening, tailored mental health literacy materials, and decision support for adolescents and/or their parents. This study will examine the effectiveness of these digital interventions using a randomized control trial with diverse community-based organizations in Kenya. In addition, the investigators will study underlying mechanisms that contribute to intervention effectiveness, as well as to use the data for precision medicine analysis (using machine learning approach). Findings will be used to improve Digital-Toolkit decision support functions and accuracy of mental health precision care.

ELIGIBILITY:
Adult parent and adolescent child will be enrolled in this study as a family.

Inclusion Criteria:

* Parent is over 18 years of age
* Parent has as an adolescent child between 11-14 years of age who attend one of our partnering schools/community-based organizations (CBOs).
* Parent is willing and able to provide consent for themselves and provide assent for their child
* Adolescent is between 11-14 years in age who attend one of our partnering schools/CBOs.
* One of adolescents adult parent (>18 years old) is "interested in" participating in this study
* Adolescent is willing and able to provide child assent

Exclusion Criteria:

* Parents (including biological and non-biological) who have no contact with adolescents for over 1 month

Ages: 11 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Universal mental health literacy scale for adolescents (UMHL-A Part A) attitude score | Baseline, Month 5
  The UMHL-A Part A consists of 8-items to assess adolescents attitude toward mental health. Each item on the measure is rated on a 5-point scale (1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; and 5=strongly agree) with a range in score from 8 to 40 with higher scores indicating a more positive attitude toward mental health.
Change in Parents Universal mental health literacy scale (UMHL) Part A attitude score | Baseline, Month 5
  The UMHL Part A consists of 8-items to assess parents attitude such as help seeking and stigma regarding mental health. Each item on the measure is rated on a 5-point scale (1=strongly disagree; 2=disagree; 3=neither agree nor disagree; 4=agree; and 5=strongly agree) with a range in score from 8 to 40 with higher scores indicating a more positive attitude toward mental health.
Change in UMHL-A Part B knowledge score | Baseline, Month 5
  The Universal mental health literacy scale for adolescents (UMHL-A) Part B consists of 9-items to assess adolescents mental health knowledge. Each item is rated on a scale (1=yes; 2=no, 0=I don't know). Scores can range from 0 to 18, higher scores indicate mental health illiteracy.
Change in Parents Universal mental health literacy scale (UMHL) Part B knowledge score | Baseline, Month 5
  The UMHL-A Part B consists of 9-items to assess parents mental health knowledge. Each item is rated on a scale (1=strongly agree; 2=disagree, 0=I don't know). Scores can range from 0 to 18, higher scores indicate mental health illiteracy.
Change in Adolescents Mental Health Literacy adapted items questionnaire score | Baseline, Month 5
  The adapted items questionnaire consists of 8-items to assess mental health knowledge. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 8 to 40 with higher scores indicating mental health literacy.
Change in parents Mental Health Literacy adapted items questionnaire score | Baseline, Month 5
  The adapted items questionnaire consists of 8-items to assess parents mental health knowledge regarding their child and family. Each item on the measure is rated on a 5-point scale (1=strongly disagree; 2=disagree; 3=undecided; 4=agree; and 5=strongly agree) with a range in score from 8 to 40 with higher scores indicating mental health literacy.
Change in Adolescents Patient-Reported Outcome Measurement Information System (PROMIS) Anxiety score (Adolescent report) | Baseline, Month 5
  The PROMIS Anxiety questionnaire consists of 8-items to assess anxiety adolescents felt within the past seven days. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 8 to 40 with higher scores indicating greater severity of anxiety.
Change in Adolescent Patient-Reported Outcome Measurement Information System (PROMIS) Anxiety score (parent report) | Baseline, Month 5
  The PROMIS Anger questionnaire consists of 8-items for parents to assess their child's behavior within the past seven days, specifically anxiety. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 8 to 40 with higher scores indicating greater severity of anxiety observed.
Change in Adolescents Patient-Reported Outcome Measurement Information System (PROMIS) Anger score (adolescent report) | Baseline, Month 5
  The PROMIS Anger questionnaire consists of 5-items to assess adolescents anger within the past seven days. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 5 to 25 with higher scores indicating greater severity of anger.
Change in Adolescent Patient-Reported Outcome Measurement Information System (PROMIS) Anger score (parent report) | Baseline, Month 5
  The PROMIS Anger questionnaire consists of 5-items for parents to assess their child's behavior within the past seven days, specifically anger. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 5 to 25 with higher scores indicating greater severity of anger observed.
Change in Adolescent Patient-Reported Outcome Measurement Information System (PROMIS) Depression score (parent report) | Baseline, Month 5
  The PROMIS Depression questionnaire consists of 6-items for parents to assess their child's behavior within the past seven days, specifically depression. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 6 to 30 with higher scores indicating greater severity of depression.
Change in Adolescents Strengths and Difficulties Questionnaire (SDQ)- S11-17 Conduct Problem Scale score (Adolescent report) | Baseline, Month 5
  The SDQ-S11-17 is a brief 5-item behavioral screening questionnaire for 11-17 year olds to assesses the impact of difficulties on the child's life. Each item is rated on a scale (0=not true; 1=somewhat true, 2=certainly true). Scores can range from 0 to 10 with higher scores indicating increased difficulties.
Change in Adolescent Strengths and Difficulties Questionnaire (SDQ) Conduct Problem Scale (10) S11-17 score (Parent report) | Baseline, Month 5
  The SDQ Conduct Problem Scale (10) S11-17 is a brief 5-item behavioral screening questionnaire for parents to assess the their child's behavior over the last six months. Each item is rated on a scale (0=not true; 1=somewhat true, 2=certainly true). Scores can range from 0-10, with higher scores indicating increased difficulties observed.
Change in Adolescent Patient Health Questionnaire (PHQ-9) score (Adolescent Report) | Baseline, Month 5
  The Patient Health Questionnaire (PHQ-9) is a self-administered version of the PRIME-MD diagnostic instrument that has been modified for teens (ages 11-17) and consists of 9 items assessing depression. Each item is rated on a scale (0=not at all; 1=several days; 2=more than half the days; 3=nearly every day). Total scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Yen Huang, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- University of Nairobi, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: keng-yen.huang@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to keng-yen.huang@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.